CLINICAL TRIAL: NCT00002303
Title: A Double-Blind, Placebo-Controlled Study With Open-Label Follow-Up To Determine the Safety and Efficacy of r-HuEPO in Patients With AIDS or Advanced ARC and Anemia
Brief Title: The Safety and Effectiveness of r-HuEPO in Patients With AIDS or Advanced AIDS-Related Complex (ARC) Who Are Anemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ortho Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 004D; H87-048
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-12

CONDITIONS: HIV Infections; Cytopenias
Keywords: Recombinant Proteins; Erythropoietin; Acquired Immunodeficiency Syndrome; Anemia; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Cytopenia; Acquired Immunodeficiency Syndrome; Anemia; AIDS-Related Complex | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
To determine the safety and efficacy of erythropoietin administered to patients with AIDS or advanced AIDS related complex ARC and anemia.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* History of any primary hematologic disease.
* Clinically significant disease / dysfunction of the pulmonary, cardiovascular, endocrine, neurologic, gastrointestinal, or genitourinary systems not attributable to underlying HIV disease.
* AIDS-related dementia.
* Uncontrolled hypertension (diastolic blood pressure > 100 mmHg).
* Presence of concomitant iron deficiency.
* Anemia attributable to factors other than AIDS or zidovudine (AZT) therapy.
* Acute opportunistic infection.
* History of seizures.

Concurrent Medication:

Excluded:

* Zidovudine (AZT) during the double-blind phase of the study.

Patients with clinically significant disease / dysfunction of the pulmonary, cardiovascular, endocrine, neurologic, gastrointestinal, or genitourinary systems not attributable to underlying AIDS are excluded.

Prior Medication:

Excluded within 30 days of study entry:

* Experimental drug or experimental device.
* Cytotoxic chemotherapy.
* Excluded within 2 months of study entry:
* Androgen therapy.
* Zidovudine (AZT) and during double-blind phase of study.

Clinical diagnosis of AIDS related anemia.

* Clinical diagnosis of AIDS or advanced AIDS related complex (ARC).
* Clinically stable for 1 month preceding study entry.

Substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Ortho Pharmaceutical Corp, Raritan, New Jersey, United States